CLINICAL TRIAL: NCT03895164
Title: Utilization of Linear Programming Approach to Develop Local Specific Food-based Complementary Feeding Recommendation for Stunting and Anemia Prevention Among Under-two Children
Brief Title: Linear Programming Approach to Develop Local Specific Food-based Complementary Feeding Recommendation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: SEAMEO Regional Centre for Food and Nutrition (Other)
Collaborators: Ministry of Health Republic of Indonesia (Unknown); Health Polytechnic of Pontianak (Unknown); Health Polytechnic of Malang (Unknown); Sambas District Health Office (Unknown); Malang District Health Office (Unknown); Indonesia University (Other)
Responsible Party: Principal Investigator, Dr.Umi Fahmida, Principal Investigator, SEAMEO Regional Centre for Food and Nutrition
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LPBadutaSM
Record Dates: First submitted 2019-01-21; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Stunting; Anemia; Complementary Feeding Recommendation; Linear Programming; Indonesia; Infant and Young Children; Problem Nutrients
MeSH Terms: conditions — Growth Disorders; Anemia

STUDY DESIGN:
Intervention Model Description: Control Group will receive standard nutrition education package from primary health care.
  Intervention Group will receive standard nutrition education package from primary health care enhanced with local specific food-based complementary feeding recommendation.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard NE (Placebo Comparator): Control Group will receive standard nutrition education package from primary health care.
  Interventions: Behavioral: Standard NE
- Enhanced NE (Experimental): Intervention Group will receive standard nutrition education package from primary health care enhanced with local specific food-based complementary feeding recommendation
  Interventions: Behavioral: Enhanced NE

INTERVENTIONS:
Behavioral: Enhanced NE — Standard nutrition education package from primary health care enhanced with local specific food-based complementary feeding recommendation
  Arms: Enhanced NE
Behavioral: Standard NE — Standard nutrition education package from primary health care
  Arms: Standard NE

SUMMARY:
Stunting and anemia amongst under-two children are attributable to poor nutrient intakes. The study evaluates the effectiveness of nutrition education on local specific food-based complementary feeding recommendation (CFR) to improve dietary patterns and nutritional intakes, as well as reduce stunting and anemia among under-two children.

ELIGIBILITY:
Inclusion Criteria:

* 6-11 months old at baseline
* living in selected area during the study
* apparently healthy
* willing to take part in the study and taken venous blood sample by getting signed consent from parents

Exclusion Criteria:

* the child does not present during venous blood sample collection

Ages: 6 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 926 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in anthropometric measurements | At baseline before intervention (week 0), at midpoint of intervention (week 12), at endpoint after intervention (week 24)
  to measure the change in length measured by using WHO growth standard length-for-Age (Z-Score) before and after intervention period.
Change in hemoglobin status | At baseline before intervention (week 0), at endpoint after intervention (week 24)
  to measure the change in hemoglobin (g/L) before and after intervention
Change in iron status | At baseline before intervention (week 0), at endpoint after intervention (week 24)
  to measure the change in serum ferritin (microgram/L) before and after intervention
Change in zinc status | At baseline before intervention (week 0), at endpoint after intervention (week 24)
  to measure the change in serum zinc (mg/L) before and after intervention

SECONDARY OUTCOMES:
Change in dietary patterns | At baseline before intervention (week 0), at midpoint of intervention (week 12), at endpoint after intervention (week 24)
  Dietary patterns will be measured by using Dietary Diversity Score
Change in iron intake | At baseline before intervention (week 0), at midpoint of intervention (week 12), at endpoint after intervention (week 24)
  iron intake (mg/day)
Change in zinc intake | At baseline before intervention (week 0), at midpoint of intervention (week 12), at endpoint after intervention (week 24)
  zinc intake (mg/day)
Change in calcium intake | At baseline before intervention (week 0), at midpoint of intervention (week 12), at endpoint after intervention (week 24)
  calcium intake (mg/day)

CONTACTS AND LOCATIONS:
Overall Officials: Umi Fahmida, Dr., Principal Investigator — SEAMEO Regional Centre for Food and Nutrition
Locations (2):
- Indonesia (2):
  - Sambas District Health Office, Sambas, West Borneo
  - Malang District Health Office, Malang, West Java